CLINICAL TRIAL: NCT05491018
Title: Creation of a Composite Indicator of Clinical and Economic Performance for French Pediatric Intensive Care Units
Brief Title: Performance for French Pediatric Intensive Care Units
Acronym: QUAL-REAPED
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Lille (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2018_98; PREPS-18-0433 (Other: DGOS number)
Record Dates: First submitted 2022-08-04; First posted 2022-08-08 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Severity of Illness Index
Keywords: Pediatric; intensive care; Severity of Illness; economic; scoring system

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Introduction. The measurement of severity scores in adult and pediatric resuscitation provides a tool for evaluating the clinical performance of resuscitation services. No pediatric studies have investigated the association between current procedure and diagnostic cost indices with pediatric ICU patient severity and mortality.

Objectives. The main objective of this project in real-life situations, in 14 French pediatric intensive care units, is to validate the recently available PIM3 and PRISM IV severity scores, which take into account the clinical dimension of performance in pediatric intensive care.

This project is a French multicenter prospective observational research project involving 14 French pediatric intensive care units belonging to the Groupe Francophone de Réanimation et Urgences Pédiatriques (GFRUP). All patients under 18 years of age admitted to the 14 pediatric intensive care units affiliated with the GFRUP and voluntarily participating in the project will be included in the study.

Expected outcomes are: Validation of PIM3 and PRISM IV scores in a French population to assess clinical performance. To develop a predictive model of mortality and a predictive model of cost in French pediatric intensive care units.

ELIGIBILITY:
Inclusion Criteria:

* All patients under 18 years of age admitted to the 14 pediatric intensive care units and voluntarily participating in the project will be included in the study.

Exclusion Criteria:

- Children of age of reason or parents/legal guardians of children refusing participation in this project will be excluded from the study.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 14 French pediatric intensive care units belonging to the Groupe Francophone de Réanimation et Urgences Pédiatriques (GFRUP)
Sampling Method: Non-Probability Sample
Enrollment: 13270 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Survival : yes / no | At PICU discharge,through study completion, an average of 2 years

SECONDARY OUTCOMES:
cost of PICU stay | At PICU discharge,through study completion, an average of 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane Leteurtre, MD,PhD, Principal Investigator — University Hospital, Lille